CLINICAL TRIAL: NCT06674265
Title: Evaluation of Safety and Efficacy Evaluation Post Intravenous Infusion of Activated NK Cells in Recurrent and Refractory High-risk Neuroblastoma Patients
Brief Title: Safety and Efficacy of Systemic Allogenic NK Cells in R/R Neuroblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Marzieh Ebrahimi (Industry)
Collaborators: Royan Institute (Other Government); Iran University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Marzieh Ebrahimi, Professor of Medical Immunology, Kian Immune Cell Company
Organization: Kian Immune Cell Company (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.ACECR.ROYAN.REC.1400.032
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Neuroblastoma, Recurrent, Refractory; Neuroblastoma (NB); Neuroblastoma in Children
Keywords: Neuroblastoma; High-Risk Neuroblastoma; Natural Killer Cell; Nk Cell; adrenal gland
MeSH Terms: conditions — Neuroblastoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Patients with refractory/recurrent neuroblastoma will receive 3 to 5 systemic injections of allogeneic NK cells during the intervals between their chemotherapy courses
  Interventions: Biological: Allogenic NK cells infusion
- Control Group (No Intervention): Patients in the control group will receive no cells and just conventional treatments will be administered to them.

INTERVENTIONS:
Biological: Allogenic NK cells infusion — Natural Killer (NK) cells are extracted from a healthy donor through apheresis and processed in a clean room using the CLINIMACS device. After quality assessment, these cells are stored at -198°C until needed. When required, the cells are thawed, washed, and evaluated for viability and sterility before being administered to the patient at a dosage of 5 × 10^6 cells per kilogram of body weight. Two further injections may be considered based on the patient's response and confirmed improvement via MRI MIBG. Injections are scheduled seven to ten days after each chemotherapy course according to the standard treatment protocol.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to assess safety and efficacy of systemic injection of allogenic NK cells in patients with refractory/recurrent high-risk neuroblastoma.

Is the injection of allogenic nk cells safe in patients with R/R high-risk neuroblastoma? Is the injection of allogenic nk cells effective in patients with R/R high-risk neuroblastoma? We will compare the NK cell administration group with a control group that receives conventional treatment to determine whether the intervention is safe and effective

DETAILED DESCRIPTION:
NK cells are isolated from healthy donors through the apheresis process and subsequently separated using the CLINIMACS device in a clean room environment. After quality assessment (sterility, viable cell count, purity, and phenotype of active cells), they are stored at -198°C until use. Upon need, the cells are thawed and washed, followed by checking their viability, count, and sterility. Children between the ages of 2 to 16 who meet the eligibility criteria will be added to the study. After admission, the cells are injected into the patient at a ratio of 5×10^6 cells per kilogram of the patient's body weight. A total of 3 injections are administered to all patients. Based on the patient's response and recovery status, the need for additional injections is evaluated. If improvements in the patient's condition are observed after the last injection and confirmed by MRI MIBG, further 2 injections can continue. The intervals between injections vary based on the patient's standard treatment, and the cells are injected 10 days after the completion of each chemotherapy course.

ELIGIBILITY:
Inclusion Criteria:

1. High-risk neuroblastoma that is resistant to standard induction therapy based on COG (Children's Oncology Group) criteria (according to INRG criteria and having received at least 4 cycles of multi-drug induction chemotherapy, and not responding to conventional treatments).
2. Evidence of relapse or progression of neuroblastoma after autologous peripheral blood stem cell transplantation or aggressive therapy.
3. A minimum life expectancy of 6 months.
4. Patients must have a pathological diagnosis of neuroblastoma and/or confirmation of tumor cells in the bone marrow with increased urinary catecholamines.
5. Measurable residual disease based on imaging findings using Curie scoring or MIBG or PET imaging criteria (1: measurable tumor of at least 10 mm in one dimension on MRI or CT scan with positive uptake on I-123 MIBG scan ("MIBG avid") oOR 2): increased FDG uptake on 18F-FDG PET-CT or PET-MRI ("PET avid")).

   -

Exclusion Criteria:

1. Insufficient bone marrow function: Platelet count > 50,000/µL, independent of transfusion (no platelet transfusion within one week). Absolute neutrophil count (ANC) maximum of 500 per microliter. Hemoglobin > 10 grams per deciliter.
2. Insufficient liver function: Plasma bilirubin level more than 1.5 times the upper limit of normal (ULN). SGPT (ALT) at least three times the upper limit of normal (a level of 45 units per liter is considered the upper limit of normal).
3. Insufficient kidney function: Creatinine clearance or estimated radioisotope GFR < 70 ml/min/1.73m². Plasma creatinine level more than 1.5 times the upper limit of normal based on age/gender.
4. Insufficient central nervous system function if seizures are present, entry into the study is not possible and if seizures are not well controlled with anticonvulsant drugs.

3- Insufficient cardiovascular function Shortening fraction < 27% by ECHO OR Ejection fraction < 50% by ECHO or gated radionuclide study.

4- Insufficient pulmonary function evidence of dyspnea at rest. Exercise intolerance. Chronic need for oxygen and room air pulse oximetry < 94% if pulse oximetry evaluation is clinically indicated. Presence of current pleural or pericardial effusion.

5- Inability to tolerate new treatment due to emergency conditions. 6- Elevated catecholamines (more than twice the ULN) or sole involvement of bone marrow (bone marrow positive for NB as the only evaluable disease without confirmatory pathology report).

7- Receiving 0.5 mg/kg/day of systemic steroids (equivalent to prednisone) for at least 7 days before enrollment.

8- Receiving CYP3A4 inducers or inhibitors at least 7 days before study enrollment.

9- Diagnosis of any other malignancy alongside the diagnosis of neuroblastoma. 10- Diarrhea > Grade 2 (4 to 6 stools per day). 11- Significant illness not covered by exclusion criteria but interfering with the study process or increasing the intensity of treatment with NK cells.

12- Participation in another clinical trial. 13- Severe impairment of major organ functions, such as renal, cardiac, hepatic, neurological, pulmonary, or gastrointestinal toxicity above Grade 2 according to the National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0 (CTC v5.0).

14- Inability to comply with protocol requirements. 15- Lack of confirmed and signed consent by the patient's guardians. 16- Evidence of HIV disease (Human Immunodeficiency Virus) or positive serology for HIV.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
NK Cell Infusion Safety | After each injection to next injection and 2 weeks after last injection
  The safety of the treatment is assessed using the Common Terminology Criteria for Adverse Events (CTCAE) checklist.

SECONDARY OUTCOMES:
Response rate comparison between control and intervention groups | 6 months and 12 months
  The response rate in patients in the control and treatment groups will be assessed and compared using MRI, MIBG, or PET scans.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Marzieh Ebrahimi, PhD. in Medical Immunology, Study Chair — Royan Institute; Dr. Mohammad Faranoush, Pediatric Oncologist, Principal Investigator — Iran University of Medical Science
Locations (1):
- Rasoul Akram Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No